CLINICAL TRIAL: NCT01335737
Title: Exercise and Inflammation: Autonomic, Affective & Cellular Mechanisms
Brief Title: Exercise and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Richard Sloan, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5948/6956R; HL094423 (Other: CU)
Record Dates: First submitted 2010-07-14; First posted 2011-04-14 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aerobic training (Experimental): 12 weeks of aerobic training, 4 times/week
  Interventions: Behavioral: aerobic training
- wait list control (Placebo Comparator): wait list control condition, 12 weeks + 4 to parallel the deconditioning protocol in active intervention group
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: aerobic training — 12 weeks of aerobic training, 4 times/week
  Other Names: Training, aerobic
  Arms: aerobic training
Behavioral: Wait list — wait list control condition
  Other Names: Condition, wait list control
  Arms: wait list control

SUMMARY:
The purpose of this study is to test the hypothesis that aerobic exercise leads to attenuation of the inflammatory response to lipopolysaccharide (LPS) stimulation.

DETAILED DESCRIPTION:
Aerobic exercise - the most widely recommended health behavior - is recognized to reduce the risk of coronary heart disease, so much so that consensus panels routinely include it as part of a cardioprotective regimen for healthy people, but the physiological or mechanistic basis of this protection is uncertain. Understanding the mechanisms has considerable public health significance because it will allow development and testing of targeted interventions to produce comparable cardioprotective effects more directly or in cases where aerobic exercise is not possible. This application proposes to test the hypothesis that aerobic training leads to attenuation of the inflammatory response to LPS stimulation and to examine the role played by exercise-induced increases in vagal activity, improvements in mood, and decreased expression of Toll Receptor 4 (TLR4), the cognate receptor for endotoxin expressed by monocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-45 years old
2. English-speaking
3. Ambulatory
4. BMI < 32
5. Pre-menopausal (women only) with regular cycle lengths between 26-32 days
6. "Average" fitness as determined by American Heart Association standards (VO2max < 43 ml/kg/min for men, < 37 ml/kg/min for women) VO2max test

Exclusion Criteria:

1. Use of anti-psychotic medications
2. Current of past major depressive disorder, or total symptom score > 10
3. BMI<18
4. Heart disease
5. Hypertension
6. Diabetes mellitus
7. Neurologic disease
8. Smoking
9. Individuals with ischemic heart disease, cardiac arrhythmias, peripheral vascular disease, orthopedic problems such as foot, leg, hip and spine problems,movement disorders, other neurological disorders affecting gait or balance, conditions or treatments associated with impaired thermoregulation, or other medical problems, for which aerobic training would be contraindicated.
10. Use of any medication with autonomic effects
11. Use of birth control medication
12. Ischemic changes, abnormal blood pressure responses, significant ectopy
13. Appears to be at high risk to be unable to adhere to study protocol

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
tumor necrosis factor (TNF-alpha) | change from before (pre) to after (post) 12 weeks of training & after 4 weeks of post-deconditioning
  TNF-alpha will be measured from whole blood samples stimulated with lipopolysaccharide

SECONDARY OUTCOMES:
Change in mood, including depressive symptomatology and negative affect | change from before (pre) to after (post) 12 weeks of training & after 4 weeks of post-deconditioning
interleukin 1 (IL-1), IL-6, IL-8, IL-10 | change from before (pre) to after (post) 12 weeks of training & after 4 weeks of post-deconditioning
  these cytokines will be measured from whole blood samples stimulated with lipopolysaccharide
TLR-4 | change from before (pre) to after (post) 12 weeks of training & after 4 weeks of post-deconditioning
  TLR-4 will be measured from blood samples
cerebral blood volume (CBV) in the dentate gyrus | change from before (pre) to after (post) 12 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Sloan, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Sloan RP, Shapiro PA, Demeersman RE, McKinley PS, Tracey KJ, Slavov I, Fang Y, Flood PD. Aerobic exercise attenuates inducible TNF production in humans. J Appl Physiol (1985). 2007 Sep;103(3):1007-11. doi: 10.1152/japplphysiol.00147.2007. Epub 2007 Jul 12. PMID 17626836
- [Derived] Sloan RP, Shapiro PA, Lauriola V, McIntyre K, Pavlicova M, Choi CJ, Choo TH, Scodes JM. The Impact of Aerobic Training on Cardiovascular Reactivity to and Recovery From Psychological and Orthostatic Challenge. Psychosom Med. 2021 Feb-Mar 01;83(2):125-137. doi: 10.1097/PSY.0000000000000896. PMID 33337592
- [Derived] McIntyre KM, Puterman E, Scodes JM, Choo TH, Choi CJ, Pavlicova M, Sloan RP. The effects of aerobic training on subclinical negative affect: A randomized controlled trial. Health Psychol. 2020 Apr;39(4):255-264. doi: 10.1037/hea0000836. Epub 2020 Jan 9. PMID 31916828